CLINICAL TRIAL: NCT03176771
Title: A Double-Blind, Randomized, Multicenter, Placebo-Controlled, Parallel, Fixed-Dose Study to Evaluate the Efficacy and Safety of MT-5199 for the Treatment in Patients With Tardive Dyskinesia (J-KINECT)
Brief Title: Efficacy and Safety of MT-5199 in Subjects With Tardive Dyskinesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-5199-J02
Record Dates: First submitted 2017-06-02; First posted 2017-06-05 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MT-5199 40 mg (Double-Blind Placebo-Controlled Period) (Experimental): MT-5199 administered as one (1) 40 mg capsule and one (1) placebo capsule, taken by mouth, every morning for 6 weeks.
  Interventions: Drug: MT-5199; Drug: Placebo
- MT-5199 80 mg (Double-Blind Placebo-Controlled Period) (Experimental): Subjects randomized to the MT-5199 80 mg dose will receive MT-5199 40 mg for the first week (administered as one (1) 40 mg capsule and one (1) placebo capsule), followed by MT-5199 80 mg administered as two (2) 40 mg capsules, taken by mouth, every morning for 5 weeks.
  Interventions: Drug: MT-5199; Drug: Placebo
- Placebo (Double-Blind Placebo-Controlled Period) (Experimental): Placebo administered as two (2) placebo capsules, taken by mouth, every morning for 6 weeks.
  Interventions: Drug: Placebo
- MT-5199 40 mg (Double-Blind Extension Period) (Experimental): At the end of Week 6, subjects will enter a double-blind extension period for 42 weeks. Subjects who were initially randomized to placebo will be re-randomized (1:1) to receive either MT-5199 40 mg or 80 mg and subjects initially randomized to MT-5199 will continue with their current dose.
  Interventions: Drug: MT-5199; Drug: Placebo
- MT-5199 80 mg (Double-Blind Extension Period) (Experimental): At the end of Week 6, subjects will enter a double-blind extension period for 42 weeks. Subjects who were initially randomized to placebo will be re-randomized (1:1) to receive either MT-5199 40 mg or 80 mg and subjects initially randomized to MT-5199 will continue with their current dose. Subjects re-randomized to receive MT-5199 80 mg will receive 40 mg for the first week.
  Interventions: Drug: MT-5199; Drug: Placebo

INTERVENTIONS:
Drug: MT-5199 — MT-5199 40 mg capsules
  Arms: MT-5199 40 mg (Double-Blind Extension Period); MT-5199 40 mg (Double-Blind Placebo-Controlled Period); MT-5199 80 mg (Double-Blind Extension Period); MT-5199 80 mg (Double-Blind Placebo-Controlled Period)
Drug: Placebo — MT-5199 placebo capsules

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MT-5199 administered once daily for the treatment of Tardive Dyskinesia (TD) symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Have one of the following clinical diagnoses for at least 3 months prior to screening: Schizophrenia or Schizoaffective Disorder, Bipolar Disorder, or Depressive Disorders.
* Have a clinical diagnosis of neuroleptic-induced TD.
* Have moderate or severe TD.
* If using maintenance medication(s) for schizophrenia or schizoaffective disorder, or bipolar disorder, or depressive disorders, be on stable doses.

Exclusion Criteria:

* Have an active, clinically significant unstable medical condition in screening period.
* Have a significant risk of suicidal or violent behavior.
* Have a known history of long QT syndrome or cardiac tachy-arrhythmia.
* Are currently pregnant or breastfeeding.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (82):
- Japan (82):
  - Aichi Psychiatric Medical Center, Aichi
  - Hotei Hospital, Aichi
  - Mikawa Hospital, Aichi
  - Okehazama Hospital Fujita Kokoro Care Center, Aichi
  - Akita City Hospital, Akita
  - Akita University Hospital, Akita
  - Hirosaki Aiseikai Hospital, Aomori
  - Minato Hospital, Aomori
  - Seinan Hospital, Aomori
  - Kohnodai Hospital , National Center for Global Health and Medicine, Chiba
  - National Hospital Organization Shimofusa Psychiatric Medical Center, Chiba
  - General incorporated association Shinkoukai Shinkouen, Ehime
  - Chikusuikai Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Hirota Clinic, Fukuoka
  - Iizukakinen Hospital, Fukuoka
  - Kuramitsu Hospital, Fukuoka
  - Minamigaoka Hospital, Fukuoka
  - Yahata Kousei Hospital, Fukuoka
  - Nanko Kokorono Clinic, Fukushima
  - Takeda General Hospital, Fukushima
  - Holy Cross Hospital, Gifu
  - Seimou Hospital, Gunma
  - Hayakawa Clinic, Hiroshima
  - Kamo Psychiatric Center, Hiroshima
  - Medical corporation KOSEIKAI KUSATSU HOSPITAL, Hiroshima
  - Mihara Hospital, Hiroshima
  - Hayashishita Hospital, Hokkaido
  - Ishikane Hospital, Hokkaido
  - National Hospital Organization Hokkaido Medical Center, Hokkaido
  - Obihiro-Kosei General Hospital, Hokkaido
  - Sapporo City General Hospital, Hokkaido
  - Teine Hospital, Hokkaido
  - Hyogo prefecture - Hyogo Mental Health Center, Hyōgo
  - Kobe University Hospital, Hyōgo
  - Medical corporation Shouhokai Toda Internal Medicine and Rehabilitation Department, Hyōgo
  - Awazu Neuropsychiatric Sanatorium, Ishikawa
  - Ishiki Hospital, Kagoshima
  - Minami Kyushu Sakura Hospital, Kagoshima
  - Taniyama Hospital, Kagoshima
  - Fujimidai Hospital, Kanagawa
  - Hatano Kosei Hospital, Kanagawa
  - Hino Hospital, Kanagawa
  - Kishiro Mental Clinic, Kanagawa
  - Kitaodawara Hospital Meihoukai Medical Corporation Association, Kanagawa
  - Shiunkai Yokohama Hospital, Kanagawa
  - Soushu Hospital, Kanagawa
  - Yatsushirokosei Hospital, Kumamoto
  - Yuge Hospital, Kumamoto
  - Sagaarashiyama Tanaka Clinic, Kyoto
  - Miyagi Psychiatric Center, Miyagi
  - Yasuda Hospital, Miyagi
  - National Hospital Organization Komoro kogen Hospital, Nagano
  - North Alps Medical Center Azumi Hospital, Nagano
  - Syonan Hospital, Nagano
  - Sanwa Central Hospital, Nagasaki
  - Nara Medical University Hospital, Nara
  - Akari Clinic, Okinawa
  - Arakaki Hospital, Okinawa
  - Samariya Hospital, Okinawa
  - Keihan Hospital, Osaka
  - Kyowakai Healthcare Corpration Hannan Hospital, Osaka
  - Hoaki Hospital, Ōita
  - Hizen Psychiatric Center, Saga
  - Rainbow & Sea Hospital, Saga
  - Sho Midori Hospital, Saitama
  - Shiga University of Medical Science Hospital, Shiga
  - Shimane University Hospital, Shimane
  - Numazu Chuo Hospital, Shizuoka
  - Abe Clinic, Tokyo
  - Hozumi Clinic, Tokyo
  - Kyorin University Hospital, Tokyo
  - Maynds Tower Mental Clinic, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
  - Nishigahara Hospital, Tokyo
  - Ongata Hospital, Tokyo
  - Sangenjaya Neurology-Psychosomatic Clinic, Tokyo
  - Senzoku Mental Clinic, Tokyo
  - Kawada Hospital, Toyama
  - Minamitoyama Nakagawa Hospital, Toyama
  - Public Okitama General Hospital, Yamagata
  - National Hospital Organization Kanmon Medical Center, Yamaguchi

REFERENCES:
- [Result] Horiguchi J, Watanabe K, Kondo K, Iwatake A, Sakamoto H, Susuta Y, Masui H, Watanabe Y. Efficacy and safety of valbenazine in Japanese patients with tardive dyskinesia: A multicenter, randomized, double-blind, placebo-controlled study (J-KINECT). Psychiatry Clin Neurosci. 2022 Nov;76(11):560-569. doi: 10.1111/pcn.13455. Epub 2022 Sep 17. PMID 36114799
- [Derived] Watanabe Y, Susuta Y, Nagano M, Masui H, Kanahara N. Efficacy and Safety of Valbenazine in Elderly and Nonelderly Japanese Patients With Tardive Dyskinesia: A Post Hoc Analysis of the J-KINECT Study. J Clin Psychopharmacol. 2024 Nov-Dec;44(6):551-560. doi: 10.1097/JCP.0000000000001903. Epub 2024 Aug 27. PMID 39186921
- [Derived] Nagano M, Susuta Y, Masui H, Watanabe Y, Watanabe K. Efficacy and Safety of Valbenazine in Japanese Patients With Tardive Dyskinesia and Schizophrenia/Schizoaffective Disorder or Bipolar Disorder/Depressive Disorder: Primary Results and Post Hoc Analyses of the J-KINECT Study. J Clin Psychopharmacol. 2024 Mar-Apr 01;44(2):107-116. doi: 10.1097/JCP.0000000000001811. PMID 38421921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled schizophrenia/schizoaffective disorder subject with tardive dyskinesia (TD), or bipolar disorder/depressive disorder with TD from 100 centers in Japan.The last patient completed in September 2020.
Groups:
- Placebo (Double-Blind Placebo-Controlled Period): Subjects who were randomized to receive Placebo capsule once daily for 6 weeks.
- MT-5199 40 mg (Double-Blind Placebo-Controlled Period): Subjects who were randomized to receive MT-5199 (Valbenazine) 40 mg capsule once daily for 6 weeks.
- MT-5199 80 mg (Double-Blind Placebo-Controlled Period): Subjects who were randomized to receive MT-5199 (Valbenazine) 40 mg capsule once daily for 1 weeks, then 80 mg capsule once daily for 5 weeks.
- MT-5199 40 mg (Double-Blind Extension Period): At the end of Week 6, subjects will enter a double-blind extension period for 42 weeks. Subjects who were initially randomized to placebo will be re-randomized (1:1) to receive either MT-5199 (Valbenazine) 40 mg or 80 mg and subjects initially randomized to MT-5199 (Valbenazine) will continue with their current dose.
- MT-5199 80 mg (Double-Blind Extension Period): At the end of Week 6, subjects will enter a double-blind extension period for 42 weeks. Subjects who were initially randomized to placebo will be re-randomized (1:1) to receive either MT-5199 (Valbenazine) 40 mg or 80 mg and subjects initially randomized to MT-5199 (Valbenazine) will continue with their current dose. Subjects re-randomized to receive MT-5199 (Valbenazine) 80 mg will receive 40 mg for the first week.
Period: Double-Blind Placebo-Controlled Period
Arm/Group | Placebo (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Extension Period) | MT-5199 80 mg (Double-Blind Extension Period)
Started | 85 | 86 | 85 | 0 | 0
Completed | 80 | 71 | 60 | 0 | 0
Not Completed | 5 | 15 | 25 | 0 | 0
Not completed — Adverse Event | 3 | 5 | 14 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 10 | 0 | 0
Not completed — Incorrect allocation | 0 | 0 | 1 | 0 | 0
Period: Double-Blind Extension Period
Arm/Group | Placebo (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Extension Period) | MT-5199 80 mg (Double-Blind Extension Period)
Started | 0 (Of the 80 placebo subjects who remained in the study at Week 6, 41 were re-randomized to MT-5199 40 mg (Double-Blind Extension Period) and 39 were re-randomized to MT-5199 80 mg (Double-Blind Extension Period).) | 0 (All MT-5199 40 mg 71 subjects who completed Double-Blind Placebo-Controlled Period entered to MT-5199 40 mg Double-Blind Extension Period.) | 0 (All MT-5199 80 mg 60 subjects who completed Double-Blind Placebo-Controlled Period entered to MT-5199 80 mg Double-Blind Extension Period.) | 112 (Of the 112 subject who entered the MT-5199 40 mg (Double-Blind Extension Period), 41 were previously in the placebo group and 71 were in the 40 mg group during the Double-Blind Placebo-Controlled Period.) | 99 (Of the 99 subjects who entered the MT-5199 80 mg (Double-Blind Extension Period), 39 were previously in the placebo group and 60 were in the 80 mg group during the Double-Blind Placebo-Controlled Period.)
Completed | 0 | 0 | 0 | 67 | 50
Not Completed | 0 | 0 | 0 | 45 | 49
Not completed — Adverse Event | 0 | 0 | 0 | 15 | 18
Not completed — Death | 0 | 0 | 0 | 3 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 24 | 26

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Groups:
- Placebo (Double-Blind Placebo-Controlled Period): Subjects received Placebo capsule (matching MT-5199 capsules) once daily for 6 weeks.
- MT-5199 40 mg (Double-Blind Placebo-Controlled Period): Subjects received MT-5199 40mg capsule once daily for 6 weeks.
- MT-5199 80 mg (Double-Blind Placebo-Controlled Period): Subjects received MT-5199 40mg capsule once daily for 1 week, then 80mg capsule once daily for 5 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period) | Total
Number analyzed (Participants) | 84 | 85 | 84 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (13.4) | 58.6 (14.0) | 58.0 (13.8) | 58.9 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 45 | 33 | 126
  Male | 36 | 40 | 51 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 84 | 85 | 84 | 253
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 84 | 85 | 84 | 253
  Non-Japanese | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score (Central Assessment) at Week 6
Description: Severity of TD symptoms assessed by AIMS dyskinesia total score (sum of items 1 through 7), as assessed by blinded central AIMS raters. The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
Time Frame: Baseline and Week 6
Population: The analysis population (80 in the placebo, 68 in the MT-5199 40 mg, and 57 in the MT-5199 80 mg) consisted of subjects who satisfy all of the following conditions:
  * Subjects in the ITT analysis set
  * Subjects for whom the Week 6 AIMS total score (central assessment) is available
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period)
Number analyzed (Participants) | 80 | 68 | 57
units on a scale | -0.1 [-0.8 to 0.5] | -2.3 [-3.0 to -1.7] | -3.7 [-4.4 to -3.0]
Statistical Analysis 1: Comparison: Placebo (Double-Blind Placebo-Controlled Period) vs MT-5199 80 mg (Double-Blind Placebo-Controlled Period); Control for multiplicity was accomplished through the a fixed-sequence testing procedure for Week 6 outcomes: * AIMS dyskinesia total score mean change from baseline (CFB): MT-5199 80 mg vs. placebo. * AIMS: MT-5199 40 mg vs. PBO. For a test result in the above list to be considered statistically significant, all of the test results higher in the list must have been significant at the 0.05 level of significance; Test type: Superiority; p < 0.001, Mixed-effect Model Repeated Measures; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-4.5 to -2.6], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Placebo (Double-Blind Placebo-Controlled Period) vs MT-5199 40 mg (Double-Blind Placebo-Controlled Period); Test type: Superiority; p < 0.001, Mixed-effect Model Repeated Measures; Median Difference (Final Values) = -2.2, 95% CI 2-sided [-3.0 to -1.3], Standard Error of Mean 0.4

2. Secondary Outcome: Percentage of Subjects With a ≥50% Improvement From Baseline in the AIMS Total Score (Central Assessment) at Week 6 (AIMS Responder)
Description: Percentage of AIMS responders (subjects who had at least a 50 percent reduction in AIMS score from baseline)
Time Frame: Week 6
Population: The analysis population (78 in the placebo, 67 in the MT-5199 40 mg, and 53 in the MT-5199 80 mg) consisted of subjects who satisfy all of the following conditions:
  * Subjects in the ITT analysis set
  * Subjects for whom the Week 6 AIMS total score (central assessment) is available and the baseline AIMS total score (central assessment) is not zero
Measure: Number; unit: percentage of AIMS responders
Arm/Group | Placebo (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period)
Number analyzed (Participants) | 78 | 67 | 53
percentage of AIMS responders | 10.3 | 23.9 | 47.2
Statistical Analysis 1: Comparison: Placebo (Double-Blind Placebo-Controlled Period) vs MT-5199 40 mg (Double-Blind Placebo-Controlled Period); Test type: Superiority; p = 0.027, Cochran-Mantel-Haenszel; Risk Difference (RD) = 13.6
Statistical Analysis 2: Comparison: Placebo (Double-Blind Placebo-Controlled Period) vs MT-5199 80 mg (Double-Blind Placebo-Controlled Period); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 36.9

3. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score (Site Assessment) at Week 6
Description: Severity of TD symptoms assessed by AIMS dyskinesia total score (sum of items 1 through 7), as assessed by blinded site AIMS raters. The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
Time Frame: Baseline and Week 6
Population: The analysis population (80 in the placebo, 68 in the MT-5199 40 mg, and 57 in the MT-5199 80 mg) consisted of subjects who satisfy all of the following conditions:
  * Subjects in the ITT analysis set
  * Subjects for whom the Week 6 AIMS total score (site assessment) is available
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period)
Number analyzed (Participants) | 80 | 68 | 57
units on a scale | -2.3 [-3.2 to -1.5] | -3.8 [-4.7 to -3.0] | -4.7 [-5.6 to -3.8]
Statistical Analysis 1: Comparison: Placebo (Double-Blind Placebo-Controlled Period) vs MT-5199 40 mg (Double-Blind Placebo-Controlled Period); Test type: Superiority; p = 0.013, Mixed-effect Model Repeated Measures; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.7 to -0.3], Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: Placebo (Double-Blind Placebo-Controlled Period) vs MT-5199 80 mg (Double-Blind Placebo-Controlled Period); Test type: Superiority; p < 0.001, Mixed-effect Model Repeated Measures; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-3.5 to -1.1], Standard Error of Mean 0.6

4. Secondary Outcome: Clinical Global Impression of Change - TD (CGI-TD) Score at Week 6
Description: Clinician's perspective of the participant's overall improvement of TD symptoms over time. The CGI-TD is based on a 7-point scale (range: 1=very much improved to 7=very much worse).
Time Frame: Week 6
Population: The analysis population (80 in the placebo, 70 in the MT-5199 40 mg, and 60 in the MT-5199 80 mg) consisted of subjects who satisfy all of the following conditions:
  * Subjects in the ITT analysis set
  * Subjects for whom the Week 6 CGI-TD score is available
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period)
Number analyzed (Participants) | 80 | 70 | 60
units on a scale | 3.4 [3.2 to 3.6] | 3.0 [2.8 to 3.3] | 2.8 [2.5 to 3.0]
Statistical Analysis 1: Comparison: Placebo (Double-Blind Placebo-Controlled Period) vs MT-5199 40 mg (Double-Blind Placebo-Controlled Period); Test type: Superiority; p = 0.021, ANOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo (Double-Blind Placebo-Controlled Period) vs MT-5199 80 mg (Double-Blind Placebo-Controlled Period); Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.0 to -0.3], Standard Error of Mean 0.2

ADVERSE EVENTS:
Time Frame: Up to Week 6 (Placebo, MT-5199 40 mg, MT-5199 80 mg), and Post Week 6 to Week 48 (MT-5199 40 mg, MT-5199 80 mg)
Description: Subjects who received Placebo or MT-5199 during each period (Double-Blind Placebo-Controlled Period* and Double-Blind Extension Period**).
  * 84 in the placebo, 85 in the MT-5199 40 mg, and 84 in the MT-5199 80 mg
  ** 108 in the MT-5199 40 mg, and 95 in the MT-5199 80 mg
Groups:
- MT-5199 40 mg (Double-Blind Placebo-Controlled Period): Subjects received MT-5199 40 mg capsule once daily for 6 weeks.
- MT-5199 80 mg (Double-Blind Placebo-Controlled Period): Subjects received MT-5199 40 mg capsule once daily for 1 week, then 80mg capsule once daily for 5 weeks.
Arm/Group | Placebo (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period) | MT-5199 40 mg (Double-Blind Extension Period) | MT-5199 80 mg (Double-Blind Extension Period)
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/85 | 0/84 | 3/108 | 4/95
Serious Adverse Events (participants affected / at risk) | 1/84 | 4/85 | 1/84 | 15/108 | 15/95
Other Adverse Events (participants affected / at risk) | 15/84 | 30/85 | 44/84 | 71/108 | 69/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-Blind Placebo-Controlled Period) (N=84) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) (N=85) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period) (N=84) | MT-5199 40 mg (Double-Blind Extension Period) (N=108) | MT-5199 80 mg (Double-Blind Extension Period) (N=95)
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Marasmus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Stupor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Panic attack (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 5 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-Blind Placebo-Controlled Period) (N=84) | MT-5199 40 mg (Double-Blind Placebo-Controlled Period) (N=85) | MT-5199 80 mg (Double-Blind Placebo-Controlled Period) (N=84) | MT-5199 40 mg (Double-Blind Extension Period) (N=108) | MT-5199 80 mg (Double-Blind Extension Period) (N=95)
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 7 | 8
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 3 | 9 | 7 | 12
Malaise (General disorders) | 0 | 5 | 4 | 5 | 6
Nasopharyngitis (Infections and infestations) | 6 | 6 | 4 | 27 | 20
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 5 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 6
Weight decreased (Investigations) | 0 | 0 | 0 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 5
Akathisia (Nervous system disorders) | 1 | 4 | 5 | 4 | 7
Dizziness (Nervous system disorders) | 1 | 0 | 3 | 4 | 5
Somnolence (Nervous system disorders) | 2 | 10 | 21 | 9 | 8
Tremor (Nervous system disorders) | 0 | 0 | 5 | 5 | 11
Anxiety (Psychiatric disorders) | 0 | 1 | 4 | 4 | 6
Depression (Psychiatric disorders) | 1 | 1 | 3 | 5 | 7
Insomnia (Psychiatric disorders) | 1 | 2 | 5 | 8 | 11
Schizophrenia (Psychiatric disorders) | 1 | 7 | 0 | 13 | 13
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT03176771/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT03176771/SAP_001.pdf